CLINICAL TRIAL: NCT01258192
Title: Multicenter,Phase ⅡStudy of Neoadjuvant Chemotherapy With Nab-paclitaxel Plus Cisplatin for Stage Ⅱ-Ⅲ Esophageal Squamous Cell Carcinoma Patients
Brief Title: Neoadjuvant Chemotherapy With Nab-paclitaxel Plus Cisplatin for Stage Ⅱ-Ⅲ Esophageal Cancer Patients
Acronym: nabPCESCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH-ESCC-01
Record Dates: First submitted 2010-12-03; First posted 2010-12-10 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; neoadjuvant chemotherapy; albumin-bound paclitaxel; cisplatin
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Albumin-Bound Paclitaxel; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel plus cisplatin (Experimental)
  Interventions: Drug: albumin-bound paclitaxel plus cisplatin

INTERVENTIONS:
Drug: albumin-bound paclitaxel plus cisplatin — neo-chemotherapy program:Albumin-bound paclitaxel:100 mg/m2, IV (in the vein) on days 1,8 of each 21 day cycle. Cisplatin 75mg/m2,IV DRIP on day 1 of each 21 day cycle.Number of Cycles: 2 cycles before operation.If it is effective ,2 cycles will be given in 6 weeks after radical resection.
  Other Names: nab-paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of neoadjuvant chemotherapy with nab-paclitaxel plus cisplatin for stage Ⅱ-Ⅲ esophageal squamous cell carcinoma patients.

DETAILED DESCRIPTION:
A surgical resection is currently the preferred treatment for esophageal cancer if the tumor is considered to be resectable without evidence of distant metastases.A higher percentage of radical resection is reported in studies using neoadjuvant chemotherapy followed by surgery versus surgery alone.The neoadjuvant chemotherapy may improve overall survival. Neoadjuvant chemotherapy with administrations of paclitaxel combined with cisplatin or carboplatin has shown effectively.Nanoparticle albumin-bound (nab)-paclitaxel has better efficacy and practically eliminates the risk of hypersensitivity reactions associated with solvent-based paclitaxel.We try to evaluate the efficacy and safety of neoadjuvant chemotherapy with nab-paclitaxel plus cisplatin for stage Ⅱ-Ⅲ esophageal squamous cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of squamous cell carcinoma of esophagus. Preoperative stage Ⅱ-Ⅲ by endoscopic ultrasound, CT of the chest and abdomen,and esophagogram.
* Age ranges from 18 to 70 years.
* Patients must not have received any prior anticancer therapy.
* Performance status of 0 to 1
* Estimated life expectancy of at least 6 months.
* Tumor can be measured according to RECIST criteria
* Signed informed consent document on file.
* Females with childbearing potential must have a negative serum pregnancy
* Adequate organ function including the following:

Bone marrow: Absolute neutrophil count (ANC) greater than or equal 1.5×109/L Platelets greater than or equal 80×109/L Haemoglobin greater than or equal 80g/L Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN), Alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN Renal: calculated creatinine clearance rate≥60ml/min. test within 7 days prior to study enrollment.

Exclusion Criteria:

* Carcinoma at the upper part of esophagus
* Histologic diagnosis of adenocarcinoma of esophagus.
* Prior treatment for esophageal cancer.
* Active infection.
* Pregnant or breast feeding.
* History of significant neurological or mental disorder, including seizures or dementia.
* Prior invasive malignancy in 5 years (except for carcinoma in situ).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
response to induction therapy | 2 years
  The response to induction therapy will be evaluated

SECONDARY OUTCOMES:
rate of complete pathological response | 2 years
  The rate of complete pathological response will be evaluated
R0 resection rate. | 2 years
  Complete resection rate to pre-operative chemotherapy will be assessed
3 years disease free and overall survival | 5 years
  Three years disease free and overall survival will be evaluated.
safety and tolerability | From time of consent to last visit
  To monitor the safety and tolerability by evaluation of the frequency, severity, and duration of treatment-emergent adverse events in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Fan Y, Jiang Y, Zhou X, Chen Q, Huang Z, Xu Y, Gong L, Yu H, Yang H, Liu J, Lei T, Zhao Q, Mao W. Phase II study of neoadjuvant therapy with nab-paclitaxel and cisplatin followed by surgery in patients with locally advanced esophageal squamous cell carcinoma. Oncotarget. 2016 Aug 2;7(31):50624-50634. doi: 10.18632/oncotarget.9562. PMID 27244882